CLINICAL TRIAL: NCT00255255
Title: An Open, Phase III, Multicentre, 52-week Study, Evaluating the Safety and Efficacy of Symbicort® Turbuhaler® (1, 2, and 4 x 160/4.5 µg Twice Daily) in Japanese Patients With Asthma
Brief Title: Safety & Efficacy of Symbicort® Turbuhaler® (1, 2, and 4 x 160/4.5 µg Twice Daily) in Japanese Patients With Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D5890C00009
Record Dates: First submitted 2005-11-17; First posted 2005-11-18 (Estimated); Last update posted 2011-01-24 (Estimated); Status verified 2011-01

CONDITIONS: Asthma
Keywords: Asthma
MeSH Terms: conditions — Asthma | interventions — Budesonide, Formoterol Fumarate Drug Combination

INTERVENTIONS:
Drug: Budesonide/Formoterol
  Other Names: Symbicort

SUMMARY:
This study is to confirm the safety of Symbicort® Turbuhaler® 160/4.5 µg 1, 2 or 4 inhalation b.i.d. over a 52 week treatment period in asthmatic patients who are being treated with IGCS and long acting β2-agonist (LABA) and/or other anti-asthmatic drugs.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of asthma with a documented history of at least 6 months duration prior to Visit 1
* Prescribed daily use of an IGCS for ≥12 weeks prior to Visit 1
* Prescribed daily use of at least one of the following:

Theophylline, long acting β2-agonist (LABA), other anti-asthmatic drugs (leucotrine antagonists, inhaled anti-cholinergics, Th2 cytokine inhibitor) for at least 4 weeks prior to Visit 1 at a constant dose

Exclusion Criteria:

* Any significant disease or disorder that may jeopardize the safety of the patient
* Respiratory infection, judged by the investigator(s) as an infection affecting the asthma, within 4 weeks prior to Visit 1
* Treatment with oral, parenteral or rectal GCS within 4 weeks prior to Visit 1

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120
Dates: Start 2005-11; Primary Completion 2006-12 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Safety: Adverse events (nature, incidence and severity) Haematology, clinical chemistry, morning plasma cortisol, urinalysis, and ACTH challenge test 12-lead ECGs, blood pressure, pulse rate

SECONDARY OUTCOMES:
Patient reported outcomes regarding disease status (incl. PEF), collected via diaries
Forced expiratory volume in one second (FEV1)
- all variables assessed over the 52 week treatment period

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Symbicort Medical Science Director, MD, Study Director — AstraZeneca
Locations (18):
- Japan (18):
  - Research Site, Komaki, Aichi-ken
  - Research Site, Seto, Aichi-ken
  - Research Site, Gifu, Gifu
  - Research Site, Ōwa, Gunma
  - Research Site, Hiroshima, Hiroshima
  - Research Site, Sapporo, Hokkaido
  - Research Site, Tomakomai, Hokkaido
  - Research Site, Morioka, Iwate
  - Research Site, Takamatsu, Kagawa-ken
  - Research Site, Kagoshima, Kagoshima-ken
  - Research Site, Kochi, Kochi
  - Research Site, Beppu, Ohita
  - Research Site, Tsukubo-gun, Okayama-ken
  - Research Site, Kishiwada, Osaka
  - Research Site, Takatsuki, Osaka
  - Research Site, Ōta-ku, Tokyo
  - Research Site, Shinjuku-ku, Tokyo
  - Research Site, Ube, Yamaguchi